CLINICAL TRIAL: NCT03450551
Title: Comparison of Clinical Efficacy of Three Class II Correctors in Orthodontics, Prospective Expertise Matched Controlled Trial
Brief Title: Comparison of Efficacy of Three Orthodontic Appliances
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108653
Record Dates: First submitted 2017-05-04; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Malocclusion, Angle Class II
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Twin Block (Experimental): 61 patients will receive the Twin Block appliance (one of the three appliances being studied)
  Interventions: Device: Twin Block, Herbst, Frog distalising appliance
- Herbst (Active Comparator): 61 patients will receive the Herbst appliance (one of the three appliances being studied)
  Interventions: Device: Twin Block, Herbst, Frog distalising appliance
- Frog distalising appliance (Active Comparator): 61 patients will receive the Frog distalising appliance (one of the three appliances being studied)
  Interventions: Device: Twin Block, Herbst, Frog distalising appliance

INTERVENTIONS:
Device: Twin Block, Herbst, Frog distalising appliance — To study which of the three orthodontic appliances does achieve the best clinical progress, produce least discomfort to the patient, minimize the time taken for completion of treatment and maximize compliance.

SUMMARY:
To investigate each treatment modality in its "optimal" environment to avoid operator experience bias. Therefore we propose to operate out of three "specialist centres" with specific units providing one modality alone Which of the three orthodontic appliances does achieve best clinical progress, produce least discomfort to the patient, minimize the time taken for completion of treatment and maximize compliance.

DETAILED DESCRIPTION:
Patients and materials: The patient population will consist of patients age 10-16 that have, or are close to having, a full permanent dentition, and present to the clinic with Class II malocclusions with more than 1/2 unit II molar relationship. (Normal or deep overbite cases are also included). The treatments to be compared are the three (routinely-used) orthodontic appliances: Twin Block, Herbst and Frog.

Hypothesis: The principal (null) hypothesis is that there is no difference between the three appliances in terms of their effectiveness, efficiency and compliance.

Study design: The study is designed as a multicentre, Prospective Expertise Based Matched Controlled Longitudinal Trial and the assessments will be longitudinal in time.

All patients that consent/assent to be part of the study (and their parents) will receive an information leaflet about the study and will be asked to sign an assent form. Patients are free to discontinue treatment if they wish to do so. The normal length of orthodontic treatment is between 18 and 24 months. Assessments will be taken prior to treatment and throughout the treatment period, with regular progress reviews every 3 months, as per standard practice.

Outcomes: The principal outcome for efficiency is the time taken for completion of treatment. The principal outcomes for effectiveness are the clinical progress, discomfort (caused by the appliance to the patient) and compliance.

Clinical progress will be assessed by measuring tooth movement on each review appointment, using radiographic examination (DPT and lateral cephalograms). Each patient will record discomfort in a visual analogue scale (VAS or Likert scale)and compliance by writing the days the appliance was not in the mouth for any reason.

Covariates: Socio-economic variables: age, gender, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 10-16 years of age in the late mixed/permanent dentition with Class II malocclusions (Both Cl II div 1 and Cl II div 2)
2. > 1/2 unit Class II molar relationship bilaterally (at least 3.5mm)
3. Normal or deep overbite cases will be included
4. Skeletal Class II relationship (ANB > 4°)
5. Overjet ≥ 5 mm in Cl II/1 cases
6. Non-extraction cases

Exclusion Criteria:

1. Children in the early mixed dentition
2. Class I and Class III malocclusions
3. Malocclusions with less than 1/2 unit II molar relationship
4. Reduced overbite / anterior openbite
5. Medically compromised patients, syndromic patients or patients with severe facial asymmetry
6. Special needs patients not able to comply with instructions / difficulty with compliance
7. Hypodontia or extracted permanent tooth (except third molars)
8. Poor oral hygiene with both Gingival bleeding Index and Plaque Index scoring no more than 1

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 183 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have experienced discomfort related to wearing the appliance | 18-24 months
  This is to check which appliance produces more discomfort compared to the other appliances using the Likert scale. Each question on the scale asks to rate the pain as either (no pain, slight pain, moderate pain, severe pain) or (strongly disagree, disagree, agree, strongly agree). Patients will choose a response which matches their experience.
establishing which appliance has the fastest completion time | 18-24 months
  The three appliances will be compared in 'months' from the start of treatment till the completion of treatment to see which is the fastest to achieve the end result

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bister, Consultant, Principal Investigator — Guy's and St Thomas NHS Trust

IPD SHARING:
Plan to Share IPD: Yes
No personal patient details will be shared. Only study data collected.